CLINICAL TRIAL: NCT00555503
Title: Registry of Mastectomy for Breast Cancer Risk Reduction
Status: Completed | Type: Observational
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, Scott L. Spear, M.D., Chief Plastic Surgery, Georgetown University
Other Study IDs: 2007-383
Record Dates: First submitted 2007-11-07; First posted 2007-11-08 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-12

CONDITIONS: Quality of Life; Mastectomy; Breast Neoplasms; Genetic Predisposition to Disease; Adjustment Disorder
Keywords: prospective study; registry; quality of life; mastectomy; reconstructive surgical procedures; BrCa1; BrCa2; breast cancer prevention
MeSH Terms: conditions — Breast Neoplasms; Genetic Predisposition to Disease; Adjustment Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patient operative specimens, blood samples, and saliva samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients who have risk-reduction mastectomy of any type, per protocol inclusion and exclusion criteria.

SUMMARY:
This is a registry for patients who have a risk-reduction mastectomy ("prophylactic mastectomy") due to being at high risk for developing breast cancer, followed by breast reconstruction. Eligible patients include those who have a breast cancer-related gene, a strong family history of breast cancer, or a personal history of high-risk conditions such as cancer in the other breast or ductal carcinoma in situ (DCIS). Patients are enrolled in the registry before surgery, and are followed for up to ten years afterwards. In addition to studying medical outcomes, we will periodically survey patients for quality-of-life issues and psychological well-being. There is no compensation for being enrolled in this registry. This registry is conducted through the Department of Plastic Surgery at Georgetown University Hospital, and is a sub-registry to the Fisher Familial Cancer Registry at the Lombardi Comprehensive Cancer Center at Georgetown University.

ELIGIBILITY:
Inclusion Criteria:

* Patients at an elevated risk for breast cancer.

Exclusion Criteria:

* None.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are enrolled from the plastic surgery, breast surgery, or oncology clinics at Georgetown University Hospital who are at elevated risk for breast cancer. Please note that the Registry can only enroll Georgetown University Hospital patients.
Sampling Method: Non-Probability Sample
Enrollment: 261 (Actual)
Dates: Start 2007-11; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
The primary study endpoint is the quality of life of the individual patient at the end of one year. Quality of life is measured using standardized self-report instruments administered preoperatively and in annual follow-up. | 10 years

SECONDARY OUTCOMES:
Cancer occurrence, adverse effects, imaging findings, and survival are all secondary outcomes that we will be following. | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Scott L. Spear, M.D., Principal Investigator — Georgetown University Hospital
Locations (1):
- Georgetown University Hospital, Washington D.C., District of Columbia, United States